CLINICAL TRIAL: NCT01566747
Title: A Phase II Study of Pazopanib in Patients With Metastatic or Unresectable Renal Cell Carcinoma (RCC) Who Have Failed Prior Sunitinib Therapy
Brief Title: Second-line Pazopanib Renal Cell Carcinoma (RCC) Study. CTRIAL-IE (ICORG) 10-01, V5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 10-01
Record Dates: First submitted 2012-03-08; First posted 2012-03-29 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

ARMS (1):
- Pazopanib (Experimental): Pazopanib 800mg day to be given continuously until disease progression.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800mg day to be given continuously until disease progression.

SUMMARY:
This is a phase II open label, single arm study evaluating treatment with pazopanib post sunitinib treatment in 43 patients with metastatic renal cell carcinoma. Patients will receive 800mg pazopanib per day given continuously until disease progression. Patients must have received treatment with sunitinib and relapsed. Patient must have received prior treatment with sunitinib for at least 12 weeks. Prior treatment with either temsirolimus or everolimus in addition to sunitinib is allowed. The trial design uses a Simons two stage design with an interim analysis planned after the first 15 evaluable patients. If 8 or more of the first 15 evaluable patients remains disease free at 4 months, then a further 28 patients will be enrolled for a total of 43 metastatic renal cell cancer patients. It is estimated that there could be up to 10% of patients dropping out and so to achieve the required number of 43 evaluable patients the study will recruit up to 48 patients to ensure that 43 complete if stage 2 is required.

Patients will receive treatment until disease progression, unacceptable toxicity or withdrawal of patient consent. Response assessments will be carried out every 8 weeks until disease progression. Safety assessments will be carried out every 4 weeks (plus a visit for liver function tests after 2 weeks) for the first six months and then every eight weeks until disease progression. A further safety assessment will be carried out 4 weeks after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.

   Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.

   Note: It is not necessary that informed consent be obtained within the protocol-specified screening window.
2. Age ≥ 18 years
3. Diagnosis of metastatic/unresectable renal cell carcinoma of the clear cell type or with a component of clear cell histology
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Measurable disease by RECIST criteria (Version 1.1)
6. Eligible patients must have been treated with sunitinib for a minimum of 12 weeks (2 cycles). Patients must have evidence of progressive disease following treatment with sunitinib as assessed by the site investigator on the basis of CT scans and other appropriate clinical documentation. Patients who received sunitinib for 12 weeks (2cycles) but stopped the drug due to toxicity rather than disease progression are also eligible for this study.

   The Investigator should be aware of the patient's intolerance/toxicity with prior sunitinib treatment and take this in to account when assessing eligibility for the pazopanib study.

   Patients who have had prior treatment with either temsirolimus or everolimus are also eligible for the trial.

   No other prior treatment with bevacizumab, sorafenib, immunotherapies, chemotherapy, biologic therapy or investigational therapy is allowed.

   Previous radiotherapy (RT) is permissible provided the measurable disease is outside the RT port. RT must be completed > 2 weeks prior to registration.
7. Adequate organ system function as defined below

   Definitions for Adequate Organ Function System Laboratory Values

   Hematologic Absolute neutrophil count (ANC) ≥ 1.5 X 109/L Hemoglobina ≥ 9 g/dL (5.6 mmol/L)

   Platelets > or = 100 X 10^9/L Prothrombin time (PT) or international normalized ratio (INR)b < or = 1.2 X ULN Activated partial thromboplastin time (aPTT) < or = 1.2 X ULN Hepatic Total bilirubin < or = 1.5 X ULN Alanine amino transferase (ALT) and Aspartate aminotransferase (AST)c < or = 2.5 X ULN Renal Serum creatinine < or = 1.5 mg/dL (133 µmol/L) Or, if >1.5 mg/dL: Calculated creatinine clearance (ClCR) (Appendix F) > or = 50 mL/min Urine Protein to Creatinine Ratio (UPC; Appendix F)d <1
   * Subjects may not have had a transfusion within 7 days of screening assessment.
   * Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
   * Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.
   * If UPC > or = 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 g to be eligible.
8. A female is eligible to enter and participate in this study if she is of:

   Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
   * A hysterectomy
   * A bilateral oophorectomy (ovariectomy)
   * A bilateral tubal ligation
   * Is post-menopausal Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).

   Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT

   Childbearing potential, including any female who has had a negative serum or urine pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
   * Oral contraceptive, either combined or progestogen alone
   * Injectable progestogen
   * Implants of levonorgestre
   * Estrogenic vaginal ring
   * Percutaneous contraceptive patches
   * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
   * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
   * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)

   Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
9. Left Ventricular Ejection Fraction > or = Lower Limit of Institutional Normal as assessed by Echocardiograph or MUGA

Exclusion criteria

1. Prior malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases (surgery plus or minus radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible: a) are asymptomatic, b) have had no evidence of active CNS metastases for > or = 6 months prior to enrolment, and c) have no requirement for steroids or Enzyme -inducing anticonvulsants EIACs.

   Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for Gastrointestinal (GI) bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with suspected bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
4. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   * Malabsorption syndrome
   * Major resection of the stomach or small bowel.
5. Presence of uncontrolled infection.
6. Prolongation of corrected QT interval (QTc) > 480 msecs using Bazett's formula
7. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) [http://www.abouthf.org/questions_stages.htm, accessed 8th December 2009]

     * Class III (Moderate): marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
     * Class IV (Severe): unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
8. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥150 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].

   Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <150/90 mmHg in order for a subject to be eligible for the study (see Appendix H for details on BP control and re-assessment prior to study enrollment).

   Note: A mean BP in 24 hours of <150/90 mm/Hg is acceptable.
9. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
10. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
11. Evidence of active bleeding or bleeding diathesis.
12. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
13. Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
14. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
15. Unable or unwilling to discontinue use of prohibited medications list in Section 6.2.4 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
16. Treatment with any of the following anti-cancer therapies:

    * Minor surgical procedure or tumor embolization within 14 days prior to the first dose of pazoapnib
    * Previous radiotherapy (RT) is permissible provided the measurable disease is outside the RT port. RT must be completed > 2 weeks prior to registration.
    * sunitinib, everolimus or temsirolimus within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib Note: No other prior treatment with bevacizumab, sorafenib, immunotherapies, chemotherapy, biologic therapy or investigational therapy is allowed.
17. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
18. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to 4 years

CONTACTS AND LOCATIONS:
Locations (9):
- Ireland (8):
  - Beaumont Hospital, Dublin, Leinster
  - Mater Misericordiae University Hospital, Dublin, Leinster
  - Mater Private Hospital, Dublin, Leinster
  - Cork University Hospital, Cork
  - The Adelaide & Meath Hospital Dublin incorporating the National Children's Hospital, Dublin
  - Galway University Hospital, Galway
  - Mid-Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford
- Karolinska University Hospital, Stockholm, Sweden